CLINICAL TRIAL: NCT07355543
Title: Prospective, Single Centre, Single-blinded, Randomized Clinical Investigation to Evaluate the Effectiveness and Safety of a Cryogenic Device to Treat Skin Tags Versus a Comparator Product.
Brief Title: Evaluate the Effectiveness and Safety of a Cryogenic Pen to Treat Skin Tags Versus a Comparator.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-0952-U5
Record Dates: First submitted 2025-11-17; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Skin Tags
Keywords: NITROFREEZE SKIN TAG; SKIN TAG

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NITROFREEZE SKIN TAG (Experimental): Topical application on the selected skin tag for 20 seconds. Maximum of 3 treatments with a 15 days interval between each treatment.
  Interventions: Device: NITROFREEZE Skin tag
- Scholl Freeze Away Skin Tag Remover (Active Comparator): Topical application on the selected skin tag for 40 seconds. Skin tag can be removed in 1 treatment. If the skin tag has not fallen off in 2 weeks, you may treat the skin tag again, up to 3 treatment cycles.
  Interventions: Device: Scholl Freeze Away Skin Tag Remover

INTERVENTIONS:
Device: NITROFREEZE Skin tag — Treatment of the skin tag with NITROFREEZE Skin Tag device on Day 0, Day 15, Day 30.
  Arms: NITROFREEZE SKIN TAG
Device: Scholl Freeze Away Skin Tag Remover — Treatment of the skin tag with Scholl Freeze Away Skin Tag Remover device on Day 0, Day 15, Day 30.
  Arms: Scholl Freeze Away Skin Tag Remover

SUMMARY:
The purpose of this clinical investigation is to evaluate the effectiveness and safety of Nitrofreeze Skin Tag for the treatment of skin tags versus a comparator device (Scholl Freeze Away® Skin Tag Remover).

DETAILED DESCRIPTION:
The primary objective of the study is to assess the efficacy of Nitrofreeze Skin Tag (tested product) for the treatment of skin tags versus a comparator product.

The secondary objectives are to assess the safety of the tested product versus comparator product.

To meet these objectives, the subjects will be monitored as follows:

At the screening visit (visit 1), the study will be explained to the subject by the investigator before any study related procedures are performed. Both the subject and the investigator will sign the consent form and the investigator will check inclusion and exclusion criteria. This can also be done at the D0 visit.

At visit 2 on D0, if the subject is eligible, the subject will perform the first treatment on the selected skin tag with the tested product or comparator, at the lab.

At visit 3 on D3, the investigator will evaluate the skin condition on and around the skin tag and collect adverse events.

At visit 4 on D15, assessment of effectiveness and safety will be made. A second treatment can be done if first treatment is not effective. Study end if the skin tag was successfully removed.

At visit 5 on D30, assessment of effectiveness and safety will be made. A third treatment can be done if second treatment is not effective. Study end if the skin tag was successfully removed.

At visit 6 on D45, assessment of effectiveness and safety will be made. Study end.

In case of missing treatment on D15 or D30 because of a missing visit or a skin condition that did not permit a new treatment, the third treatment will be done on D45. In that case, a new follow-up visit will be done at D60.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject.
2. Sex: male or female.
3. Age: more than 22 years old.
4. Phototype: I to III according to Fitzpatrick.
5. Subject presenting at least one skin tag that could be treated by the tested devices as evaluated by the investigator:

   * Location: on the neck, chest, back, groin or underarm;
   * Colour: skin tags must be similar in colour to the surrounding skin;
   * Shape & Feel: skin tags must be soft and flexible.
   * Size: 2 to 5 mm in size.
6. Subject having given freely and expressly his/her informed consent.
7. Subject who is able to comply with the study requirements, as defined in the present CIP, at the investigator's appreciation.
8. Subject affiliated to a health social security system.
9. Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before screening visit and during all the study.

Exclusion Criteria:

1. Pregnant or nursing woman or planning a pregnancy during the study.
2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
3. Subject in a social or sanitary establishment.
4. Subject having received 6000 euros indemnities for participation in clinical research in the 12 previous months, including participation in the present study.
5. Subject enrolled in another clinical trial or which exclusion period is not over.
6. Member of the CRO or the centre staff.
7. Subject with a condition or receiving a medication which, in the investigator's judgment, put the subject at undue risk.
8. Subject suffering from a severe or progressive disease (including asthma and diabetes).
9. Subject with immune deficiency or autoimmune disease.
10. Subject suffering from an acute or cutaneous disease or any other cutaneous pathology.
11. Subject with a history of skin cancer or pre-cancerous skin lesions.
12. Subject with previous event of healing disorders such as hypertrophic or keloid scar, residual pigmentation etc.
13. Subject with blood circulation or blood clotting problems including Raynaud's disease; blood dyscrasias of unknown origin; haemophilia subjects.
14. Subject presenting skin growths such as birthmarks, moles, warts, or any other unusual-looking skin condition on the treated zone.
15. Subject having thin, inflamed, damaged, irritated, itchy, infected, cut, grazed, diseased or red skin on and around the treated zone.
16. Subject with molluscum contagiosum, blisters or any other vesicles on the skin on and around the treated zone.
17. Subject with a known allergy to Chlorhexidine based antiseptic or to adhesives.
18. Subject who already had an abnormal reaction to cold.
19. Subject whose selected skin tag is bleeding or scratched.
20. Subject whose skin tag is located on the face, scalp or mucosa, anus, genitals, buttocks, lips, eyelids or eyes.
21. Subject undergoing a topical treatment on the test area or a systemic treatment:

    * anti-inflammatory medication within 5 days prior to D0 visit,
    * immunosuppressors and/or corticoids within 10 days prior to D0 visit,
    * retinoids within 6 months prior to D0 visit,
    * treatment with an action on coagulation within 1 week prior to D0 visit,
    * any long-term medication stabilized for less than one month.
22. Subject who received a treatment of any kind on the selected skin tag within 6 months prior to D0 visit.
23. Intensive exposure to sunlight or UV-rays within the previous month and/or foreseen exposure of the treated zone during the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate | From enrollment to the end of treatment at 60 days (maximum)
  Comparison of the percentage of subjects having a successful treatment of the selected skin tag in the Nitrofreeze Skin Tag group versus comparator group by clinical evaluation by the blinded evaluator.
  The investigator, who will be in blind of the treatment administered, will measure the selected skin tag height and diameter in mm before treatment on day 0, day 3, day 15, day 30, day 45 and day 60 if applicable.
  At each timepoint after first treatment session, the blinded investigator will rate the treatment success using the following scale:
  0= No change
  1. Improvement
  2. Disappearance of skin tag
  The percentage of subjects having a successful treatment at study end will be calculated for the investigational device and comparator. The treatment is considered successful if the blinded investigator scores the selected skin tag as "2".
  If the score is evaluated as 0 or 1 at a follow-up visit, a new treatment will be done (maximum 3 treatments).

SECONDARY OUTCOMES:
Global effectiveness-subjective questionnaire | Study end (day 15, day 30, day 45 or day 60 according to the treatment success)
  A subjective evaluation questionnaire, will be filled in by the subjects at study end to evaluate the devices global effectiveness. This questionnaire contains 18 questions concerning effectiveness, where the subjects can score the device with "Agree", "Somewhat Agree", "Neither agree nor disagree", "Disagree" or "Not applicable"
Skin condition | From enrollment to the end of the treatment at 60 days (maximum)
  Evaluation of the skin condition at each timepoint by clinical evaluation by the blinded investigator.
  The investigator will evaluate the clinical signs observed on the skin tag and on the healthy skin surrounding the skin tag before treatment on day 0, day 3, day 15, day 30, day 45 and day 60 if applicable using the following clinical scores:
  * None (0)
  * Mild (1)
  * Moderate (2)
  * Severe (3)
Pain during treatment by the subject | From enrollment to the end of treatment at 60 days (maximum)
  The subjects will be asked to evaluate the pain felt during each treatment on a visual analogic scale of 10 cm.
Pain and healing process by the subject | From enrolment to the end of treatment at 60 days (maximum)
  The subjects will score every day until next visit in their daily diary the following signs: pain (scale: none, mild, moderate, severe) as well as redness, black colour, blister, wound and scab (scale: absence, presence) in order to evaluate the healing process. The subjects will also be asked to write down any other intolerance reactions that have occurred during the study in the diary.
Global tolerability | Study end (Day 15, Day 30, Day 45 or Day 60 according to the treatment success)
  According to the signs observed at each timepoint, the global tolerability of the investigational device and comparator will be defined by the blinded investigator on the following scale at the study end:
  0= Bad tolerance:
  1. Moderate tolerance
  2. Good tolerance
  3. Very good tolerance.
Amount and severity of Adverse Events (AEs) | From enrolment to the end of treatment at 60 days (maximum)
  General tolerance by collection of amount and severity of Adverse Events (AEs) by the blinded investigator for the whole study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan Pharmascan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No